CLINICAL TRIAL: NCT01158235
Title: A Randomised, Double-blind, Placebo-controlled, Ascending Dose Phase I/IIa Study to Evaluate the Safety, Tolerability and Efficacy of Topical LTX-109 in Subjects Nasally Colonized With Methicillin-resistant/-Sensitive Staphylococcus Aureus (MRSA/MSSA)
Brief Title: A Phase I/IIa Study to Evaluate the Safety, Tolerability and Efficacy of Topical LTX-109 in Subjects Nasally Colonized With Methicillin-resistant/-Sensitive Staphylococcus Aureus (MRSA/MSSA)
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Lytix Biopharma AS (Industry)
Responsible Party: Wenche Marie Olsen, Director of Development, Infectious Diseases, Lytix Biopharma AS
Allocation: Randomized | Model: Single Group | Masking: Triple
Other Study IDs: C10-109-02
Record Dates: First submitted 2010-07-07; First posted 2010-07-08 (Estimated); Last update posted 2011-06-08 (Estimated); Status verified 2011-06

CONDITIONS: Nasal Carriers MRSA
Keywords: MRSA; nose
MeSH Terms: interventions — L-arginyl-2,5,7-tris(1,1-dimethylethyl)-L-tryptophyl-N-(2-phenylethyl)-L-argininamide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- LTX-109 (Lytixar) (Experimental): Ascending dose study. Start enrollment to group 1: 1% LTX-109/placebo, then group 2: 2%LTX-109/placebo and finally group 3: 5%LTX-109/placebo dosed in each nostril TID for 3 consecutive days.
  Interventions: Drug: LTX-109

INTERVENTIONS:
Drug: LTX-109 — 1%, 2% and 3% Lytixar (gel formulation). TID for 3 days.
  Other Names: Lytixar

SUMMARY:
This is a pilot study conducted to evaluate the safety, local tolerability and efficacy of LTX-109(Lytixar™), a lytic peptide designed to kill bacterias quickly and efficient. LTX-109 (Lytixar™)will be applied in the anterior nares in subjects who are carriers of nasal colonies of MRSA/MSSA.

The extent of systemic absorption of LTX -109 when applied to the anterior nares will be evaluated and the effect of Lytixar™ as to clear colonies of MRSA/MSSA during the the observation period and Week 2 to Week 9 after treatment.

DETAILED DESCRIPTION:
Subjects with persistent colonies of MRSA/MSSA in the nostril will be recruited to receive either active treatment or placebo. This is a dose escalating study. First grout will receive either 1% Lytixar™ or placebo, next group 2% Lytixar™ or placebo and finally 5% Lytixar™ or placebo. Dose escalation will be performed after a brief safety evaluation of the tolerability after application of Lytixar™/placebo vehicle TID for three days. Pharmacokinetic samples will be collected from subjects who are willing. Subjects will be followed until 9 weeks after initiation of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects between the ages of 16 and 75, inclusive.
* Female subjects must be non-pregnant, non-lactating.
* Female subjects of child bearing potential and male subjects with female partners of child-bearing potential must use an adequate form of diaphragm or condom with spermicidal prior to entry into the study and two weeks following the completion of all follow-up procedures 9 weeks after treatment. Hormone contraception or hormonal IUDs alone are not acceptable contraception
* Signed and dated written informed consent by subject.
* Subject's medical condition is stable, with no clinically significant abnormalities.
* Subject's pre-study laboratory screen of haematology, clinical chemistry and urinalysis are normal or if abnormal, not considered clinically significant.
* Subjects must be able to understand the subject information and the consent form, and be willing to return to the study site for follow up visits, comply with requirements, instructions and restrictions of the study listed in the informed consent form.
* All family members, to a subject carrying MRSA (not applicable for MSSA positive) should also be screened for MRSA. Subjects that are eligible may be included in the study, and family members not eligible or willing to participate should be offered treatment for decolonization of MRSA according to standard treatment and investigators choice.

Exclusion Criteria:

* Negative nasal culture for MRSA/MSSA on the first screen visit.
* Negative nasal cultures for MRSA/MSSA at any occasion during the run-in period day -14 to -3 day prior to Baseline.
* Severe eczema (eczema infected with MRSA) or skin wounds, clinically significant according to investigator.
* Previous or concurrent treatment with antimicrobials for an infection within the last 28 days prior to baseline.
* MRSA decolonization attempt in the previous 6 months (prior treatment for a MRSA infection is not an exclusion criterion).
* Systolic BP is ≥170 mmHg, or diastolic BP is ≥100 mmHg or HR is ≥110 bpm.
* Inability to take medications nasally.
* Evidence of active rhinitis, sinusitis, or upper respiratory infection.
* Disease in the region of the application sites, significant history of trauma or skin disease in the region of the application sites, current nasal skin or nasal septum condition requiring treatment or nasal surgery in the previous 3 months.
* Significant ongoing or history of drug or alcohol abuse in the opinion of the investigator makes the subject unsuitable for enrolment.
* Use of prescription or non prescription drugs within minimum 7 days prior to the first dose of study medication. Subjects on stable doses of non-prescription painkillers, anti-inflammatory drugs (such as paracetamol and NSAIDs), oral antidiabetics or insulin may be allowed to be included to the study at the discretion of the investigator.
* Known allergic reactions or hypersensitivity of significant severity in general and specifically to any component of the study medication.
* Systemic illness requiring treatment within 28 days prior to baseline.
* Clinically significant illness (defined by the investigator) in the past 4 weeks before the Screening visit.
* Current or history of significant hepatic, renal, endocrine, cardiac, nervous, psychiatric, gastrointestinal, pulmonary, haematological, or metabolic disorder that is not in a stable condition. Malignancy <5 years since final treatment.
* Current or history of any significant disease or condition known to interfere with the absorption, distribution, metabolism or excretion of drugs.
* Known positive test for Human Immunodeficiency Virus (HIV) antibody, hepatitis B virus surface antigen or hepatitis C virus antibody.
* Other unspecified reasons that, in the opinion of the investigator make the subject unsuitable for enrolment.
* Treatment with an investigational drug within 30 days prior to the first dose of study medication.

Ages: 16 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2010-05; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
Local tolerability in the anterior nares | Day 1, 2, 3. week 2-9 after final treatment.
  To explore safety, local tolerability and efficacy of LTX-109 when applied topically into the anterior nares in subjects with nasal colonisation of MRSA/MSSA. To determine the extent of systemic absorption of LTX -109 when applied to the anterior nares.

SECONDARY OUTCOMES:
To evaluate recurrence of MRSA/MSSA during the observation period. | Week 2 to Week 9 after treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Anna Nilsson, MD, PhD, Principal Investigator — Skåne University hospital, Malmö
Locations (1):
- Skåne University Hospital, Malmo, Sweden

REFERENCES:
- [Derived] Nilsson AC, Janson H, Wold H, Fugelli A, Andersson K, Hakangard C, Olsson P, Olsen WM. LTX-109 is a novel agent for nasal decolonization of methicillin-resistant and -sensitive Staphylococcus aureus. Antimicrob Agents Chemother. 2015 Jan;59(1):145-51. doi: 10.1128/AAC.03513-14. Epub 2014 Oct 20. PMID 25331699